CLINICAL TRIAL: NCT03656900
Title: Monocentric Pilot Study, for a Randomized, Crossover, Blinded Trial: Comparison of the Therapeutic Efficacy of Low Frequency Repeated Transcranial Magnetic Stimulation on Cortical Area 9 Compared to Brodmann Area 46 in the Treatment of Depressive Disorders.
Acronym: rTMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TROJAK 2009
Record Dates: First submitted 2018-08-31; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Patients With Resistant Depressive Disorders
MeSH Terms: interventions — Independent Medical Evaluation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BA9/BA46 (Experimental)
  Interventions: Device: rTMS BA9/BA46; Radiation: brain MRI; Other: Medical evaluation; Other: Psychological assessment
- BA46/BA9 (Experimental)
  Interventions: Device: rTMS BA46/BA9; Radiation: brain MRI; Other: Medical evaluation; Other: Psychological assessment

INTERVENTIONS:
Device: rTMS BA9/BA46 — 10 sessions of low-frequency repeated transcranial magnetic stimulation over two weeks on cortical area 9, then 4 weeks wash-out, then 10 sessions of low-frequency repeated transcranial magnetic stimulation repeated low frequency over two weeks on cortical area 46.
  Arms: BA9/BA46
Device: rTMS BA46/BA9 — 10 sessions of low-frequency repeated transcranial magnetic stimulation over two weeks on cortical area 46, then 4 weeks wash-out, then 10 sessions of low-frequency repeated transcranial magnetic stimulation repeated low frequency over two weeks on cortical area 9.
  Arms: BA46/BA9
Radiation: brain MRI — T1 weighted full-head high-resolution MRI with 1 mm seam cuts and sagittal orientation.
Other: Medical evaluation — complete evaluation with 6 scales (HDRS, MADRS, Beck, CGI, COVI, UKU)
Other: Psychological assessment — Subjective Life Profile Assessment (SLPA) and Helping Alliance Assessment

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a new therapeutic tool used in psychiatry. Non-invasive, well tolerated and requiring no premedication, it is performed on an outpatient basis. The principle of this technique is to stimulate the cerebral cortex from an electromagnetic coil placed on the scalp. Unlike electroconvulsive therapy, rTMS induces an electrical current on a well-defined region of the cerebral cortex.

In psychiatry, this technique is mainly considered in the treatment of depressive disorders resistant to antidepressant medication. The brain target, obtained from brain imaging data in depressed patients, is the dorsolateral prefrontal cortex (DLPFC). The Food and Drug Administration (FDA) has recognized the interest of rTMS for treating depressive disorders (October 7, 2008).

However, some stimulation parameters still need to be optimized before rTMS can be considered a therapeutic method in its own right and used routinely. Indeed, its effectiveness over time has not yet been evaluated, and rTMS has shown a lack of reproducibility between subjects [Foucher, 2007]. Finally, the therapeutic results of rTMS are very modest whatever the study [Daskalakis, 2008]. Additional studies are therefore needed to optimize stimulation parameters.

ELIGIBILITY:
Inclusion Criteria:

Patients with resistant depressive disorders (Hamilton-17-item scale > 22, failure ≥ 2 antidepressants) with at least one of the following criteria :

* venlafaxine treatment failure (unlike the national PHRC, patients who receive/have received venlafaxine treatment for the current depressive episode are included),
* therapeutic failure in PHRC national rTMS 2007,
* refusal to participate in the PHRC national rTMS 2007.

Exclusion Criteria:

* Bipolar disorders: type I or II,
* Depression with psychotic characteristics,
* Schizophrenia,
* Risky or harmful use of alcohol and/or an illicit psychoactive substance,
* Dependence on alcohol and/or an illicit psychoactive substance,
* Sick and hospitalized under duress or under legal protection (guardianship, curatorship),
* Contraindication to the practice of rTMS; personal history of seizures, history of neurological or neurosurgical pathologies, metallic prosthetic materials or foreign bodies (pacemaker, etc...),
* Contraindication to brain MRI,
* Pregnancy or breastfeeding in progress
* Resistance to Escitalopram

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The remission rate | Through study completion, an average of 11 weeks.
  Compare the remission rates (decrease < 50% of the HDRS score / initial score) during neuronavigated stimulations on BA 9 and BA 46 compared to the average rate obtained during manual stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France